CLINICAL TRIAL: NCT04266145
Title: Intravenous Versus Perineural Dexmedetomidine as Adjuvant in Adductor Canal Block for Total Knee Arthroplasty
Acronym: dexmed_ACB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: dexmedetomidine
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Post Spinal Anesthesia Shivering
Keywords: dexmedetomidine-adductor canal block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study anesthetic drugs both for adductor-canal-blockade and for intravenous infusion were prepared according to the group by an anesthetist who was not involved in its injection or the perioperative assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous dexmedetomidine (Active Comparator): 20 mL 0.25% levobupivacaine plus 1 mL normal saline will be administrated for adductor-canal-blockade while for intravenous solution; 0.5µg.kg-1 dexmedetomidine diluted in 20 mL normal saline will be prepared
  Interventions: Drug: intravenous dexmedetomidine
- adductor-canal-blockade dexmedetomidine (Active Comparator): 20 mL 0.25% levobupivacaine containing 1 mL of 0.5 mcg.kg-1 dexmedetomidine will be used for adductor-canal-blockade whereas, 20 mL 0.9% saline will be prepared for intravenous infusion
  Interventions: Drug: adductor canal block dexmedetomidine

INTERVENTIONS:
Drug: intravenous dexmedetomidine — adductor-canal-blockade with 20 mL 0.25% levobupivacaine plus 1 mL normal saline while, the intravenous solution; consists of 0.5µg.kg-1 dexmedetomidine diluted in 20 mL normal saline
  Arms: intravenous dexmedetomidine
Drug: adductor canal block dexmedetomidine — adductor-canal-blockade with 20 mL 0.25% levobupivacaine plus 1 mL of 0.5µg.kg-1 dexmedetomidineline while, the intravenous solution;consists of 20 mL normal saline
  Arms: adductor-canal-blockade dexmedetomidine

SUMMARY:
Shivering increases the cardiac and systemic energy expenditure, oxygen consumption and carbon dioxide production. Definitive prevention and treatment of shivering is necessary to decrease the related complications and increase post-anesthetic comfort.

DETAILED DESCRIPTION:
Dexmedetomidine a highly selective α2 adrenergic agonist used effectively as a safe analgesic via different routes and mechanisms, including intravenous (i.v.), neuraxial and perineural routes. Dexmedetomidine has been used for prevent shivering but, the results of its efficacy is still controversy.

No studies to date have investigated the best administration route of dexmedetomidine to dominantly prevent the occurrence of shivering after spinal anesthesia or associated with the least grade.

This prospective, randomized, double blinded study was designed to investigate the best administrative route of dexmedetomidine firstly, as a preventive of neuraxial shivering and secondly as adjunctive analgesic.

The incidence of post-spinal anesthesia shivering was the primary outcome. Perioperative hemodynamics, postoperative pain scores during rest and at 45-degree flexion of the knee, the analgesic duration, the first postoperative day analgesic consumption, the sedation score and early ambulation ability were the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* both genders
* American Society of Anesthesiologists physical status I and II
* scheduled for unilateral primary TKA under spinal anesthesia

Exclusion Criteria:

* chronic opioid use
* known allergy to the used drugs
* any contraindications to regional anesthesia like; patient refusal, coagulopathy, neuropathy or infection at the injection site

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-02-29 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
incidence of post-spinal anesthesia shivering | up to 24 hours
  5-point scale (0= no shivering, 1 =piloerection or peripheral vasoconstriction but no visible shivering; 2 =muscular activity in only one muscle group; 3 =muscular activity in more than one muscle group but not generalized and 4 = shivering involving the whole body)

SECONDARY OUTCOMES:
The analgesic duration | during the first postoperative 24 hours
  the time from adductor-canal-blockade injection till the first of postoperative dose of rescue analgesic
total cumulative doses of rescue analgesic | after the first postoperative 24 hours
  given when visual analog scale for pain ≥ 40
Modified Ramsay sedation scale | after 0.5 hour from adductor-canal-blockade then, 2, 4, 6, 8, 10, 12 and 24 hours postoperatively
  1. Awake and alert, minimal or no cognitive impairment
  2. Awake but tranquil, purposeful responses to verbal commands at a conversational level
  3. Appears asleep, purposeful response to verbal commands at a conversational level
  4. Appears asleep, purposeful responses to commands but at a louder than conversational level, requiring light glabellar tap, or both
  5. Asleep, sluggish purposeful responses only to loud verbal commands, strong glabellar tap, or both
  6. Asleep, sluggish purposeful responses only to painful stimuli
  7. Asleep, reflex withdrawal to painful stimuli only
  8. Unresponsive to external stimuli, including pain
non-invasive arterial blood pressure | every 15 minutes after spinal anesthesia till the end of the surgery then at 0.5, 1, 3, 6, 12 hours postoperative
  mmHg
Heart rate | every 15 minutes after spinal anesthesia till the end of the surgery then at 0.5, 1, 3, 6, 12 hours postoperative
  beat per minute
postoperative pain | preoperative, 2, 4, 6, 8, 10, 12 and 24 hours postoperatively
  visual analog scale for pain (0 mm= no pain, and 100 = the worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Abozeid, MD, Principal Investigator — Faculty of Medicine - Mansoura University
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Egypt